CLINICAL TRIAL: NCT01402960
Title: Exploration of Parameters of tDCS in Chronic Pain Patients
Brief Title: Exploration of Parameters of Transcranial Direct Current Stimulation (tDCS) in Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Felipe Fregni, Principal Investigator, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Device Feasibility
Other Study IDs: 2010-p-000990
Record Dates: First submitted 2011-06-29; First posted 2011-07-26 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Chronic Pain
Keywords: High-Definition Transcranial Direct Current Stimulation
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (3):
- Active Anodal HD-tDCS (Experimental): Subject will receive one 20-minute session of active anodal HD-tDCS.
  Interventions: Device: High Definition Transcranial Direct Current Stimulation (HD-tDCS)
- Active Cathodal HD-tDCS (Experimental): Subject will receive one 20-minute session of active cathodal HD-tDCS.
  Interventions: Device: High Definition Transcranial Direct Current Stimulation (HD-tDCS)
- Sham HD-tDCS (Sham Comparator): Subject will receive one sham session of HD-tDCS
  Interventions: Device: High Definition Transcranial Direct Current Stimulation (HD-tDCS)

INTERVENTIONS:
Device: High Definition Transcranial Direct Current Stimulation (HD-tDCS) — Subject will receive active anodal/cathodal and sham HD-tDCS in a randomized, counterbalanced order. Each stimulation session will be separated by at least one week to avoid carryover effects. For both active and sham HD-tDCS the electrodes will be placed over the primary motor cortex, at an intensity of 2mA.
  * For active anodal stimulation, the anode will be over the primary motor cortex, and the cathodal electrodes (4) will surround the anode in a 3 inch square, duration will be 20 minutes.
  * For active cathodal stimulation, the cathode will be over the primary motor cortex, and the anodal electrodes (4) will surround the cathode in a 3 inch square, duration will be 20 minutes.
  * For sham stimulation, the same procedure will be used, however, current will only be active for 30 seconds (current ramping up, then ramping down)

SUMMARY:
The purpose of this study is to assess the effects of high-definition transcranial direct current stimulation (HD-tDCS) on subjects with chronic musculoskeletal pain. The investigators hypothesize that subjects will show a decrease in pain symptoms in the active anodal stimulation group when compared to sham stimulation.

ELIGIBILITY:
STUDY ELIGIBILITY CRITERIA

Inclusion Criteria:

1. Providing informed consent to participate in the study
2. 18 to 64 years old
3. Having chronic musculoskeletal pain (existing pain for more than 6 months with an average of at least 3 on a 0-10 VAS scale)
4. Pain resistant to common analgesics and medications for chronic pain such as Tylenol, Aspirin, Ibuprofen, Soma, Parafon Forte DCS, Zanaflex, and Codeine.
5. Must have the ability to feel pain as self reported

Exclusion Criteria:

1. Pregnancy
2. Contraindications to tDCS

   * metal in the head
   * implanted brain medical devices
3. History of alcohol or drug abuse within the past 6 months as self reported
4. Use of carbamazepine within the past 6 months as self reported.
5. Severe depression (with a score of >30 in the Beck Depression Inventory)
6. History of neurological disorders as self reported.
7. History of unexplained fainting spells as self reported,
8. History of head injury resulting in more than a momentary loss of consciousness as self reported
9. History of neurosurgery as self reported

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2011-04; Primary Completion 2012-02 (Actual); Study Completion 2013-02-13 (Actual)

PRIMARY OUTCOMES:
Change in pain scales | Measured for approximately 5 weeks
  Determine whether anodal or cathodal hd-tDCS is effective in reducing pain in subjects with chronic musculoskeletal pain as measured by changes in the Visual Analogue Scale (VAS) for pain. The VAS scale will be measured immediately before the hd-tDCS stimulation sessions and after the hd-tDCS stimulation sessions for each subject for the duration of their participation in the trial. This outcome will also be measured at their baseline visit, and follow-up visit.

SECONDARY OUTCOMES:
Change in cutaneous hyperalgesia/allodynia | Measured for approximately 5 weeks.
  To investigate whether treatment with active anodal hd-tDCS alters the phenomenon of central sensitization as indexed by cutaneous allodynia and hyperalgesia by measuring whether anodal tDCS changes the threshold for pain and perception as compared with sham and cathodal hd-tDCS. The subject's pain threshold will be measured immediately before the hd-tDCS stimulation sessions and after the hd-tDCS stimulation sessions for the duration of their participation in the trial. This outcome will also be measured at their baseline visit, and follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Fregni, MD, PhD, MPH, Principal Investigator — Spaulding Rehabilitation Hospital (SRH)
Locations (1):
- Spaulding Rehabilitation Hospital, Boston, Massachusetts, United States